CLINICAL TRIAL: NCT02789969
Title: A Randomized Controlled Trial to Compare Pain Medications in Children Undergoing Strabismus Surgery
Brief Title: Pain Medications in Children Undergoing Strabismus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Louis Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201602156
Record Dates: First submitted 2016-05-23; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Pain; Nausea
MeSH Terms: conditions — Pain; Nausea | interventions — Hydromorphone; Fentanyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydromorphone 15mcg/kg IV (Experimental): Patient randomly assigned to hydromorphone
  Interventions: Drug: Hydromorphone
- Fentanyl 1.5 mcg/kg IV (Experimental): Patient randomly assigned to fentanyl
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Hydromorphone — Hydromorphone 15mcg/kg IV
  Other Names: Dilaudid
  Arms: Hydromorphone 15mcg/kg IV
Drug: Fentanyl — Fentanyl 1.5mcg/kg IV
  Other Names: Sublimaze
  Arms: Fentanyl 1.5 mcg/kg IV

SUMMARY:
Every year over 1,000 children undergo eye muscle surgery provided by physicians at this institution. For many of these children this is not and will not be the only surgical procedure for eye muscle correction. All of these children will experience differing degrees of postoperative pain. The pain associated with strabismus surgery is due to the manipulation in the conjunctival area and further handling of Tenon's capsule, sclera and the stretching of the eye muscle . Research has demonstrated that repeated painful procedures result in increased anxiety and increased pain.

Previous studies have demonstrated that children experiencing preoperative anxiety are more likely to have increased postoperative pain . This increased preoperative anxiety may also contribute to sleep difficulties and increased analgesic consumption. Depending on the age of the child, different methods are used to reduce anxiety such as distraction, child life services, or anti-anxiolytic agents.

In addition to pain, children undergoing strabismus surgery frequently experience postoperative nausea and vomiting (PONV).This increased incidence of nausea and vomiting is thought to be related to the use of opiates for pain control. Short acting opiates are used preferentially at this hospital in the belief that this reduces recovery issues of sedation and PONV. Preliminary data, however, suggests no difference in recovery outcomes for fentanyl versus hydromorphone. The purpose of this study is to investigate the optimal analgesia to create a standardized approach for pain management in pediatric patients undergoing surgery for strabismus.

DETAILED DESCRIPTION:
Research Design This is a randomized clinical trial with masked assessment, comparing recovery indices for patients receiving longer acting versus shorter acting opiate analgesia using hydromorphone or fentanyl as intraoperative analgesics. An otherwise standardized anesthetic and analgesic regimen will be utilized, as consistent with routine care at the research institution.

Sample and Setting Patients included will be children age 3 through 10 years scheduled for strabismus surgery. The procedure may also include scheduled exam under anesthesia (EUA) of the eyes, but any other surgical procedure in conjunction with strabismus will be excluded from enrollment. Review of anesthesia records shows that 480 patients met inclusion criteria for the preceding 12 months. The primary outcome measure is pain as measured by the revised Faces, Legs, Anxiety, Cry & Consolability scale (rFLACC). Based on previous pilot work, the investigators expect pain scores to have a mean of five and a standard deviation of two. The goal is to detect a change of one point in rFLACC scores, which the investigators believe would be clinically significant. With alpha of 0.05 and power of 0.80, the investigators would need 64 patients in each arm for a one point decrease in rFLACC scores to be statistically significant. The investigators expect that ten percent of patients will have to be dropped because of missing data, so the investigators are proposing to enroll 71 patients in each arm (142 patients total) in order to have data for 64 patients in the analyses.

Inclusion criteria will be 1) children ages 3 to 10 years old having strabismus surgery for the first time, a repeated strabismus surgery, or an eye examination for strabismus under anesthesia; 2) the child has to be evaluated as an American Society of Anesthesiologists Physical Status (ASAPS) classification Class 1 or 2; 3) the caregiver should be present in the hospital; and 4) the child and caregiver must be English speaking. Exclusion criteria will include 1) children evaluated as an ASAPS Class 3 or 4; non-English speaking children or parents; 3) additional surgery performed at the same time; 4) children with documented behavioral disabilities; 5) prior participation in the study.

Tools A researcher developed demographic questionnaire will be used to collect information from a parent that includes patient age, gender, previous surgery, any medication allergies, and primary caregiver. The Amsterdam Preoperative Anxiety and Information Scale (APAIS) will be used to assess parent feelings of anxiety in the preoperative phase. The APAIS is short 6-item questionnaire with acceptable reliability with Cronbach's alpha greater than or equal to 70 and correlated highly (0.74) with the widely used State Trait Anxiety Scale. Because of its length, the APAIS can be quickly administered to parents of children undergoing surgery in order to assess parental preoperative anxiety . The measure will be completed on all parent participants after consent is obtained. The tool takes approximately 1-2 minutes to score.

For evaluating anxiety in children the Modified Anxiety Scale (mYPAS) will be used. The mYPAS is frequently used to measure anxiety prior to induction and has demonstrated both inter and intra-rater reliability (using k statistics) ranging from 0.63 - 0.90 and acceptable reliability (p = 0.01, r = 0.79) The tool can be administered in less than one minute, is reliable in children ages 2-12 years, and uses five areas (activity, vocalization, expression, arousal, and interaction) to rate preoperative anxiety.

In the Post Anesthesia Care Unit (PACU) and in Same Day Surgery (SDS), nurses will use the rFLACC scale to measure pain. The tool has established reliability and validity and is used throughout the hospital to assess pain in children unable to verbalize pain. The interrater reliability revealed intra-class correlation coefficients ranging from 0.76-0.90. Criterion validity (p=0.65-0.87) was supported by correlations between parent and child scores. For pain assessment at 24 hours post operatively, parents will be asked to rate the intensity of the subject's pain on a scale of 0 (no pain) to 10 (worst pain imaginable). The Numeric Pain Rating Scale developed by McCaffery is a widely used instrument in the clinical setting with previously established reliability and validity. The instrument is scored as 0 = no pain; 1-3 = mild pain; 4-6 = moderate pain; 7-10 = severe pain.

Procedure IRB approval will be secured prior to recruitment. As is standard care, subjects will be contacted by telephone in the days prior to the scheduled surgery. During that contact, subjects will be informed of the offer to participate in this study, and be provided with a brief description of the protocol. On the day of surgery, a researcher will visit interested subjects and provide a complete explanation and written consent document.

Consenting subjects will then be evaluated with the Amsterdam Preoperative Anxiety Scale, and the researcher will complete the YPAS-m scale prior to surgery. At the time consent is obtained, subjects will also be asked to complete a brief demographic data form.

After surgery, the nurse will evaluate the patient's pain using rFLACC scale on arrival to the Post Anesthesia Care Unit (PACU) and every fifteen minutes during the patient's stay. After transferring from PACU to SDS, the nurse will continue to evaluate pain using the same scale on arrival and before discharge. The nurse will document the patient's level of pain and need for any additional pain medication. To help ensure study fidelity in regard to pain assessment, all nurses will be given a refresher class on use of the rFLACC. After discharge, the patient will receive a telephone call 24 hours after surgery to evaluate post-operative nausea and vomiting and the level of pain at home.

Patients will receive a standard anesthetic consisting of midazolam premedication when indicated for anticipated separation anxiety, then sevoflurane inhalation utilizing nitrous oxide during mask induction, but no nitrous oxide during maintenance anesthesia. Analgesia and PONV prophylaxis is standardized as acetaminophen 15 mg/kg oral preoperative (maximum 650), followed by ketorolac 0.5 mg/kg IV (maximum 30), ondansetron 0.15 mg/kg IV, and dexamethasone 0.15 mg/kg IV. Airway maintenance will be with a laryngeal mask, and emergence conducted in the operating room with the aim of a responsive patient at time of departure from the operating room.

Patients will be randomized to either hydromorphone or fentanyl once in the operating room by opening a sealed protocol envelope. The anesthesiologist will fractionate the total dose opiate administered as the clinical situation warrants to preserve spontaneous breathing. The anesthesiologist will titrate the same drug as required during the first 15 minutes in the recovery room to ensure that immediate analgesic goals are met.

ELIGIBILITY:
Inclusion Criteria:

* ages 3 to 10 years old having strabismus surgery for the first time, a repeated strabismus surgery, or an eye examination for strabismus under anesthesia;
* evaluated as an American Society of Anesthesiologists Physical Status (ASAPS) classification Class 1 or 2
* the caregiver should be present in the hospital
* the child and caregiver must be English speaking.

Exclusion Criteria:

* evaluated as an ASAPS Class 3 or 4
* non-English speaking children or parents
* additional surgery performed at the same time
* documented behavioral disabilities
* prior participation in the study.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change in pain measured by the rFLACC scale | every 15 minutes for 2 hours and 24 hours after discharge

SECONDARY OUTCOMES:
nausea measured by self-report | every 15 minutes for 2 hours and 24 hours after discharge
Parental anxiety measured by Amsterdam Preoperative Anxiety and Information Scale | 1 time preoperatively 1 hour before surgery
  patient anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Hasima Hajdini, BSN, Principal Investigator — St. Louis Children's Hospital; Charles Schrock, MD, Study Director — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noel M, McMurtry CM, Chambers CT, McGrath PJ. Children's memory for painful procedures: the relationship of pain intensity, anxiety, and adult behaviors to subsequent recall. J Pediatr Psychol. 2010 Jul;35(6):626-36. doi: 10.1093/jpepsy/jsp096. Epub 2009 Nov 4. PMID 19889718
- [Background] Bakr RH, Abdelaziz HM. SUBTENON BUPIVACAINE INJECTION FOR POSTOPERATIVE PAIN RELIEF FOLLOWING PEDIATRIC STRABISMUS SURGERY: A RANDOMIZED CONTROLLED DOUBLE BLIND TRIAL. Middle East J Anaesthesiol. 2015 Feb;23(1):91-9. PMID 26121900
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Chieng YJ, Chan WC, Klainin-Yobas P, He HG. Perioperative anxiety and postoperative pain in children and adolescents undergoing elective surgical procedures: a quantitative systematic review. J Adv Nurs. 2014 Feb;70(2):243-55. doi: 10.1111/jan.12205. Epub 2013 Jul 19. PMID 23865442
- [Background] Chieng YJ, Chan WC, Liam JL, Klainin-Yobas P, Wang W, He HG. Exploring influencing factors of postoperative pain in school-age children undergoing elective surgery. J Spec Pediatr Nurs. 2013 Jul;18(3):243-52. doi: 10.1111/jspn.12030. Epub 2013 Apr 23. PMID 23822848
- [Background] Brasher C, Gafsous B, Dugue S, Thiollier A, Kinderf J, Nivoche Y, Grace R, Dahmani S. Postoperative pain management in children and infants: an update. Paediatr Drugs. 2014 Apr;16(2):129-40. doi: 10.1007/s40272-013-0062-0. PMID 24407716
- [Background] He HG, Zhu L, Chan SW, Klainin-Yobas P, Wang W. The effectiveness of therapeutic play intervention in reducing perioperative anxiety, negative behaviors, and postoperative pain in children undergoing elective surgery: a systematic review. Pain Manag Nurs. 2015 Jun;16(3):425-39. doi: 10.1016/j.pmn.2014.08.011. PMID 26025800
- [Background] He HG, Zhu L, Li HC, Wang W, Vehvilainen-Julkunen K, Chan SW. A randomized controlled trial of the effectiveness of a therapeutic play intervention on outcomes of children undergoing inpatient elective surgery: study protocol. J Adv Nurs. 2014 Feb;70(2):431-42. doi: 10.1111/jan.12234. Epub 2013 Aug 29. PMID 23991679
- [Background] Chhabra A, Pandey R, Khandelwal M, Subramaniam R, Gupta S. Anesthetic techniques and postoperative emesis in pediatric strabismus surgery. Reg Anesth Pain Med. 2005 Jan-Feb;30(1):43-7. doi: 10.1016/j.rapm.2004.08.023. PMID 15690267